CLINICAL TRIAL: NCT02372617
Title: Hip Reconstruction in Cerebral Palsy With Pelvic Osteotomy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Associação de Assistência a Criança Deficiente (Other)
Responsible Party: Principal Investigator, Mauro Cesar de Morais Filho, Chief of Orthopedic Staff, Associação de Assistência a Criança Deficiente
Other Study IDs: AACD 30/2011
Record Dates: First submitted 2015-02-22; First posted 2015-02-26 (Estimated); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Cerebral Palsy
Keywords: cerebral palsy; hip; luxation; subluxation
MeSH Terms: conditions — Cerebral Palsy; Joint Dislocations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group A: bone graft - autologous
  Interventions: Procedure: periacetabular osteotomy
- Group B: bone graft - ceramic
  Interventions: Procedure: periacetabular osteotomy

INTERVENTIONS:
Procedure: periacetabular osteotomy

SUMMARY:
Prospective study enrolling patients with cerebral palsy and with subluxation of the hips > 40% and acetabular dysplasia. The patients will be stratified according the degree of subluxation and age. The treatment protocol is composed by femur variation osteotomy and periacetabular osteotomy. Patients will be divided in two groups according the type of bone graft used at periacetabular osteotomy (autologous or ceramic).

ELIGIBILITY:
Inclusion Criteria:

* hip subluxation > 40% and acetabular dysplasia

Exclusion Criteria:

* previous hip surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with cerebral palsy of AACD Cerebral Palsy Clinic, with progressive hip subluxation.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Acetabular index | 12 months

SECONDARY OUTCOMES:
Reimers Index | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- AACD, São Paulo, São Paulo, Brazil